CLINICAL TRIAL: NCT07216053
Title: Predictive Value of Lung Ultrasound for Respiratory Decompensation in Late Preterm Neonates
Status: Recruiting | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: Pro2025-0102
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Pre-Term; Respiratory Distress of Newborn; Premature
Keywords: Lung Ultrasound; Respiratory Decompensation; Late Preterm Neonates; respiratory distress
MeSH Terms: conditions — Premature Birth; Pulmonary Atelectasis; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Point of care lung ultrasound: Recruited babies will undergo point-of-care lung ultrasound (POC LUS) in their first 4 hours of life and be scored based on three established scoring systems. Infants will be followed during initial hospitalization. Respiratory decompensation will be determined by 48 hours of life. If respiratory decompensation occurs, the onset of signs of respiratory distress (determined by initiation of respiratory support) and the severity of respiratory distress (determined by length of time on respiratory support) will be measured.
  Interventions: Diagnostic Test: Point of care lung ultrasound

INTERVENTIONS:
Diagnostic Test: Point of care lung ultrasound — Point-of-care lung ultrasound (POC LUS) in their first 4 hours of life and be scored based on three established scoring systems

SUMMARY:
Respiratory morbidity presents a significant clinical challenge in the neonatal period, and an individual patient's clinical course is often difficult to predict. This is especially true for late-preterm infants, who share some of the same risks of premature babies in terms or respiratory morbidity, but whose births may not always be attended by a neonatologist, or who may be born at hospitals with lower level Neonatal Intensive Care Units (NICUs) and require transfer if they decompensate.

With this study, the aim is to 1) determine the efficacy of early point of care lung ultrasound (LUS) to predict respiratory decompensation in the first 48 hours of life in late preterm infants and 2) to compare the performance of three lung ultrasound scoring systems, 3 type-of-lung, high risk pattern and total LUS scoring systems.

DETAILED DESCRIPTION:
Respiratory morbidity presents a significant clinical challenge in the neonatal period, and an individual patient's clinical course is often difficult to predict. This is especially true for late-preterm infants, who share some of the same risks of premature babies in terms or respiratory morbidity, but whose births may not always be attended by a neonatologist, or who may be born at hospitals with lower level Neonatal Intensive Care Units (NICUs) and require transfer if they decompensate.

Point of care (POC) lung ultrasound (LUS) is a relatively new and potentially underused method of assessing a neonate's respiratory status. The imaging modality has long been used to assess for common pulmonary pathologies such as pleural effusion and pneumothorax, but recent studies have begun to examine the utility of POC LUS for predicting a patient's clinical course, and potential need for escalation of respiratory support or NICU admission.

Existing studies regarding POC LUS as a predictor of need for respiratory support have focused primarily on either extremely or moderately premature or term infants, showing that three different scoring systems have been effective in predicting need for future respiratory support. Some studies have included late preterm infants, but this population reflected only a small portion of total study participants, and others did not include them at all. Given that late preterm neonates are a unique and at-risk population, the paucity of data in the existing knowledge presents a gap that should be addressed.

This study proposes conducting a prospective observational study that focuses on late preterm infants, which will assess whether the existing POC LUS scoring methodologies are useful in this population and will compare the efficacy of these scoring systems. It is proposed to recruit any infant born in the late preterm period who is initially on room air (RA) or nasal cannula (NC), conducting POC LUS and assigning scores per each of the three scoring systems, and assessing their respective predictive values for respiratory decompensation/escalation of support.

ELIGIBILITY:
Inclusion Criteria:

* Inborn infants born between 34w0d and 36w6d gestational age
* In RA or 1 Litre per minute 1LPM NC (room air (RA) or nasal cannula (NC))
* Admitted to NICU or Well Baby Nursery (WBN)

Exclusion Criteria:

* Patients born <34 weeks or >36w6d
* Major genetic anomaly or syndromic condition
* Cardiac or pulmonary structural defects
* Cord pH <7.0 or 5 minute APGAR 5 or less
* Suspected fetal hemorrhage or other source of significant anemia at birth

Ages: 34 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Inborn infants born between 34w0d and 36w6d gestational age are admitted to the NICU or Well Baby Nursery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy of POC LUS scoring systems to predict respiratory decompensation in late preterm infants. | Initial POC LUS will be performed within the first 4 hours of life. Escalation of respiratory support determined in the first 48 hours of life.
  The binary outcome of escalation vs non-escalation of respiratory support will be used to predict the accuracy of the three established POC LUS scoring systems (Three type-of-lung, Full LUS, high-risk pattern assessment) for identifying late preterm infants who experience respiratory decompensation. Respiration decompensation is defined by need for respiratory support in the form of HFNC (high flow nasal cannula), CPAP (continuous positive airway pressure), NIMV (non-invasive mechanical ventilation), mechanical ventilation or surfactant administration in infants initially in room air (RA) or nasal cannula (NC). Sensitivity, specificity, and area under ROC curve can be used to calculate the predictive accuracy. Escalation of respiratory support determined in the first 48 hours of life.
Compare the predictive accuracy of the three scoring systems | Initial POC LUS will be performed within the first 4 hours of life. Escalation of respiratory support determined in the first 48 hours of life.
  Comparison of the three POC LUS scoring systems performed in the first 4 hours of life to determine accuracy in predicting respiratory decompensation in the first 48 hours of life in late preterm infants. All three scores will be compared to the ultrasound results.

SECONDARY OUTCOMES:
Correlation between POC LUS and the timing of signs of respiratory distress | Initial POCl LUS will be performed within the first 4 hours of life. Respiratory decompensation will be determined in the first 48 hours of life.
  Determine if severity of POC LUS score correlates with onset of respiratory decompensation (i.e. does a worse LUS score correlate with earlier onset of respiratory decompensation).
Correlation between POC LUS and the severity of respiratory distress as determined by the length of support needed. | Initial POCl LUS will be performed within the first 4 hours of life. Respiratory decompensation will be determined in the first 48 hours of life.
  Determine if severity of POC LUS score correlates with the length of time infant requires respiratory support in the form of HFNC, CPAP, NIMV or mechanical ventilation (i.e. does a worse LUS score correlate with earlier onset of respiratory decompensation).
Correlation between POC LUS and the severity of respiratory distress as determined by the need for invasive respiratory support. | Initial POCl LUS will be performed within the first 4 hours of life. Respiratory decompensation will be determined in the first 48 hours of life.
  Determine if severity of POC LUS score correlates with the need for invasive versus non-invasive respiratory support.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Spillane, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Univeristy Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raimondi F, Migliaro F, Sodano A, Ferrara T, Lama S, Vallone G, Capasso L. Use of neonatal chest ultrasound to predict noninvasive ventilation failure. Pediatrics. 2014 Oct;134(4):e1089-94. doi: 10.1542/peds.2013-3924. Epub 2014 Sep 1. PMID 25180278
- [Background] Poerio A, Galletti S, Baldazzi M, Martini S, Rollo A, Spinedi S, Raimondi F, Zompatori M, Corvaglia L, Aceti A. Lung ultrasound features predict admission to the neonatal intensive care unit in infants with transient neonatal tachypnoea or respiratory distress syndrome born by caesarean section. Eur J Pediatr. 2021 Mar;180(3):869-876. doi: 10.1007/s00431-020-03789-z. Epub 2020 Sep 19. PMID 32949291
- [Background] Xi G, Dai J, Wang X, Luo F, Lu C, Yang Y, Wang J. Ultrasound performed shortly after birth can predict the respiratory support needs of late preterm and term infants: A diagnostic accuracy study. Pediatr Pulmonol. 2021 Jul;56(7):2155-2163. doi: 10.1002/ppul.25389. Epub 2021 Apr 12. PMID 33768734
- [Background] Brat R, Yousef N, Klifa R, Reynaud S, Shankar Aguilera S, De Luca D. Lung Ultrasonography Score to Evaluate Oxygenation and Surfactant Need in Neonates Treated With Continuous Positive Airway Pressure. JAMA Pediatr. 2015 Aug;169(8):e151797. doi: 10.1001/jamapediatrics.2015.1797. Epub 2015 Aug 3. PMID 26237465
- [Background] Carnazzo SM, Nasikas S, Comisi FF. Lung Ultrasound in Neonates: A Narrative Review Along With Diagnostic Insights and Early Postnatal Applications. Cureus. 2024 Sep 30;16(9):e70487. doi: 10.7759/cureus.70487. eCollection 2024 Sep. PMID 39479113